CLINICAL TRIAL: NCT02553577
Title: The Impact of Electronic Cigarettes on Perinatal Immune Responsiveness and Birth Outcomes in Appalachia
Brief Title: Impact of Electronic Cigarettes on Perinatal Immune Responsiveness and Birth Outcomes
Status: Completed | Type: Observational
Sponsor: Kristin Ashford (Other)
Collaborators: Virginia Commonwealth University (Other)
Responsible Party: Sponsor-Investigator, Kristin Ashford, Principal Investigator, University of Kentucky
Organization: University of Kentucky (Other)
Other Study IDs: 1R01DA040694-01 (NIH)
Record Dates: First submitted 2015-09-04; First posted 2015-09-17 (Estimated); Last update posted 2021-07-07 (Actual); Status verified 2021-07

CONDITIONS: Immune Response; Birth Weight; Gestational Age
Keywords: prenatal; cytokines
MeSH Terms: conditions — Birth Weight

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum cytokines: interleukin (IL) IL-1α, IL1β, IL-6, IL-8, IL-10, CRP, TNFα and MMP-8 Urinary Cotinine Urinary ( NNAL) 4-(methylnitrosamino)-1-(3-pyridyl)-1-butanone (NNK) and its metabolite 4-(methylnitrosamino)-1-(3-pyridyl)-1-butanol Expired Carbon Monoxide
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Conventional cigarettes -only: Women who are pregnant and use conventional tobacco products -only
- Electronic Cigarette (ecig) (ENDS) -ONLY: Women who are pregnant and use electronic cigarettes (ecigs) -only
- Conventional + ecig use (DUAL): Women who are pregnant and use conventional + ecigs (dual)

SUMMARY:
There has been a dramatic escalation of electronic cigarette (e-cig) use among women of childbearing age, including pregnant women. The overall goal of this study is to determine the effects of e-cigs on prenatal biomarkers and birth outcomes. It is imperative that more data about these effects be available to better inform women of childbearing age.

DETAILED DESCRIPTION:
The United States has the largest and fastest growing market for electronic cigarettes (e-cigs), and adult women of childbearing age are the most common users. However, no data exist regarding the health effects of e-cigs on pregnant women or their babies. It is well known that tobacco use during pregnancy is the most modifiable risk associated with adverse birth outcome, yet nearly one in four women in Kentucky continue to use tobacco products during pregnancy. E-cigs also contain varied (unregulated) concentrations of nicotine, despite nicotine being classified as a pregnancy class-D drug (exhibiting teratogenic effects on the fetus). The addictive nature of nicotine may explain continued use during this vulnerable time.

E-cigs have been the center of recent controversy regarding novel smoking cessation or harm reduction products. There is also concern that marketing strategies promoting harm reduction may increase the appeal and obfuscate the known adverse effects of nicotine on fetal development. In addition to the adverse effects of prenatal nicotine, maternal tobacco use alters immune response during pregnancy, placing women at increased risk for preterm birth.

The overall goal of this study is to determine the effects of e-cigs (and dual use) on perinatal biomarkers and birth outcomes. Three hundred and sixty pregnant women will be recruited. Participants will complete a survey to measure tobacco related behaviors, and provide perinatal biomarkers at four time points (each trimester and postpartum). Data analysis will include a series of repeated ANCOVAs to determine the association of perinatal cigarette smoking (conventional, e-cigarettes-only, and dual use) with perinatal biomarkers. A one-way ANCOVA will be used to determine the association with birth outcomes. Primary biomarker measures include: expired air carbon monoxide, urine and serum cotinine, serum immune markers and urinary NNAL. Gestational age at birth and birth weight are the primary birth outcomes.

Until more data about the effects of e-cigs and dual use on perinatal immune response and birth outcomes are available, promotion of e-cigs during pregnancy would be premature. There is an urgent need to investigate the impact of e-cigs and dual use on perinatal biomarkers and birth outcomes. The lack of research may unnecessarily place women-and their babies -at risk for lifelong adverse health outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. current tobacco use (traditional cigarettes and/or electronic cigarettes ecig, ENDS)
2. pregnant in the first or second trimester
3. age 18-44
4. can read and write in English.

Exclusion Criteria:

-

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant and postpartum women, age 18-44 who use tobacco products (traditional cigarettes, ENDS, electronic cigarettes)
Sampling Method: Non-Probability Sample
Enrollment: 278 (Actual)
Dates: Start 2016-01-13 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Gestational age at birth | Up to nine months
  Investigators will determine if there is a significant difference in gestational age at birth among three groups: pregnant women who use conventional tobacco-only; pregnant women who use e-cig only; and dual users

SECONDARY OUTCOMES:
Infant birth weight | Up to two hours
  Investigators will determine if there is a significant difference in birth weight among three groups: pregnant women who use conventional tobacco-only; pregnant women who use e-cig only; and dual users
Change in Prenatal Cytokine level in each trimester and postpartum | 14 weeks; 24 weeks; 34 weeks; 48 weeks and up to 64 weeks
  Investigators will determine if there are significant changes in cytokine level between trimesters based on groups hree groups: pregnant women who use conventional tobacco-only; pregnant women who use e-cig only; and dual users

CONTACTS AND LOCATIONS:
Overall Officials: Kristin B Ashford, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky Prenatal Clinics, Good Samaritian and Polk Dalton, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No